CLINICAL TRIAL: NCT01129362
Title: Surveillance for Rates of Pertussis Disease Among Persons Birth Through 59 Months of Age Receiving Pentacel® or Other Pertussis Vaccines
Brief Title: Rates of Pertussis Disease Among Persons Receiving Pentacel® or Other Pertussis Vaccines
Status: Completed | Type: Observational
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Other Study IDs: M5A16; UTN: U1111-1111-5171 (Other: WHO); NCT01079039 (obsolete NCT alias)
Record Dates: First submitted 2010-05-20; First posted 2010-05-24 (Estimated); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Pertussis
Keywords: Pertussis; Whooping Cough; Pertussis Vaccine
MeSH Terms: conditions — Whooping Cough | interventions — pentacel; diphtheria-tetanus-five component acellular pertussis-inactivated poliomyelitis -Haemophilus influenzae type b conjugate vaccine; Diphtheria-Tetanus-acellular Pertussis Vaccines; diphtheria-tetanus-pertussis-haemophilus b conjugate vaccine; PEDIARIX

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Group 1: Participants that only received Pentacel® vaccine.
  Interventions: Biological: Pentacel® (DTaP-IPV/Hib)
- Group 2: Participants that only received a single brand of pertussis vaccine other than Pentacel® vaccine.
  Interventions: Biological: Other Pertussis Vaccines
- Group 3: Participants that received more than one brand of Pertussis vaccine or one or more doses of an unknown brand.
  Interventions: Biological: Other Pertussis Vaccines

INTERVENTIONS:
Biological: Pentacel® (DTaP-IPV/Hib) — 0.5 mL dose, Intramuscular
  Other Names: Pentacel®
  Groups: Group 1
Biological: Other Pertussis Vaccines — 0.5 mL, Intramuscular
  Other Names: DAPTACEL®; Tripedia®; TriHIBit®; Infanrix®; Pediarix®
  Groups: Group 2; Group 3

SUMMARY:
The purpose of this cohort study is to determine vaccine-specific rates of pertussis disease during the period of the study, among Wisconsin residents younger than 60 months of age (the Surveillance Population), and to descriptively compare the proportion of such persons vaccinated with Pentacel® vaccine who acquire pertussis disease to the proportion of such persons vaccinated with any other Diphtheria and Tetanus Toxoids and Acellular Pertussis (DTaP) vaccine who acquire pertussis disease.

Primary Objective:

To determine the rates and relative risk of pertussis disease among Surveillance Population members who have received Pentacel vaccine or another pertussis vaccine.

DETAILED DESCRIPTION:
The study will be conducted by the University of Wisconsin School of Medicine and Public Health, in collaboration with the Wisconsin Division of Public Health (WDPH).

Epidemiological and laboratory surveillance for pertussis disease among Wisconsin residents is routinely conducted by the WDPH. During the period of the study, de-identified data regarding all incident pertussis cases will be obtained from WDPH and vaccination coverage rates, by vaccine regimen, age group, and period of time, will be obtained from ongoing marketplace surveillance conducted on behalf of the Sponsor by a national sample-survey organization. Using these data, rates of pertussis disease will be determined.

No vaccine will be administered as part of this study.

ELIGIBILITY:
Inclusion Criteria :

* Persons will be under surveillance for this study whenever the following three conditions are true: the individual resides in Wisconsin, is age birth through 59 months, and is within the surveillance period of 01 October 2009 through 30 September 2014 (or as extended in order to accrue 61,761 person years of Pentacel vaccine exposure).

Exclusion Criteria :

* Not applicable

Max Age: 59 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Wisconsin residents younger than 60 months of age.
Sampling Method: Non-Probability Sample
Enrollment: 1195 (Actual)
Dates: Start 2010-02-08 (Actual); Primary Completion 2014-12-30 (Actual); Study Completion 2014-12-30 (Actual)

PRIMARY OUTCOMES:
Occurrence of pertussis disease, as determined by the Wisconsin Division of Public Health (WDPH) | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur Inc.
Locations (1):
- Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Conway JH, Davis JP, Eickhoff JC, Pool V, Greenberg DP, Decker MD. Brand-specific rates of pertussis disease among Wisconsin children given 1-4 doses of pertussis Vaccine, 2010-2014. Vaccine. 2020 Oct 21;38(45):7063-7069. doi: 10.1016/j.vaccine.2020.09.016. Epub 2020 Sep 11. PMID 32921507
- [Derived] Decker MD, Hosbach P, Johnson DR, Pool V, Greenberg DP. Estimating the effectiveness of tetanus-diphtheria-acellular pertussis vaccine. J Infect Dis. 2015 Feb 1;211(3):497-8. doi: 10.1093/infdis/jiu477. Epub 2014 Aug 25. No abstract available. PMID 25156560